CLINICAL TRIAL: NCT07226128
Title: A Randomized, Controlled Trial Assessing the Effects of Cognitive Behavioral Therapy to Prevent Worsening Insulin Resistance in Depressed, Virologically-Suppressed, Antiretroviral-Treated Adults With HIV
Brief Title: The Effects of Cognitive Behavioral Therapy on Insulin Resistance in People With HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Samir K. Gupta, MD, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28855; R01DK141366 (NIH)
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: HIV; Depression in Adults; Insulin Resistance; Cognitive Behavior Therapy
Keywords: hiv; depression; insulin resistance; diabetes; cognitive behavioral therapy
MeSH Terms: conditions — Insulin Resistance; Acquired Immunodeficiency Syndrome; Depression; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Cognitive Behavioral Therapy (iCBT-D) (Experimental): Intervention participants will receive the empirically supported, HIPAA-compliant, therapist-assisted iCBT-D called Good Days Ahead (GDA; MindStreet, Inc.).
  GDA uses an interactive, multimedia format (including video, exercises, calls to action, newsfeeds, and customized feedback) to deliver nine 45-minute sessions, the structure and content of which mirror traditional face-to-face CBT. Topics include identifying and modifying automatic thoughts, using behavioral activation and other behavioral methods, identifying and modifying schemas, using effective coping strategies, and employing other core CBT methods.
  Interventions: Behavioral: Internet cognitive behavioral therapy (iCBT-D)
- Active Control (AC) (Active Comparator): Our AC comparator will include depression education and depressive symptom monitoring along with usual depression care as provided by the participants HIV clinicians. Trial staff will fist have a 30-minute call with AC participants to review depression materials, including their HIV provider's role in its management and treatment options and also provide a list of local mental health services. There are no care restrictions by the primary HIV clinicians. Trial staff will call AC participants every 4 weeks to assess depressive symptoms (PHQ-9) and will notify clinic staff to encourage additional care when indicated.
  Interventions: Behavioral: Active Control (AC)

INTERVENTIONS:
Behavioral: Internet cognitive behavioral therapy (iCBT-D) — Intervention participants will receive the empirically supported, HIPAA-compliant, therapist-assisted iCBT-D called Good Days Ahead (GDA; MindStreet, Inc.). GDA uses an interactive, multimedia format (including video, exercises, calls to action, newsfeeds, and customized feedback) to deliver nine 45-minute sessions, the structure and content of which mirror traditional face-to-face CBT. Topics include identifying and modifying automatic thoughts, using behavioral activation and other behavioral methods, identifying and modifying schemas, using effective coping strategies, and employing other core CBT methods.
  Arms: Internet Cognitive Behavioral Therapy (iCBT-D)
Behavioral: Active Control (AC) — Our AC comparator will include depression education and depressive symptom monitoring along with usual depression care as provided by the participants HIV clinicians. Trial staff will fist have a 30-minute call with AC participants to review depression materials, including their HIV provider's role in its management and treatment options and also provide a list of local mental health services. There are no care restrictions by the primary HIV clinicians. Trial staff will call AC participants every 4 weeks to assess depressive symptoms (PHQ-9) and will notify clinic staff to encourage additional care when indicated.
  Arms: Active Control (AC)

SUMMARY:
The goal of this clinical trial is to learn if depression treatment improves insulin resistance, or how the body uses insulin to lower blood sugar, in people with HIV on HIV treatment. Researchers will compare an internet-based (online) depression treatment program called cognitive behavioral therapy with depression education. In the online group, participants will undergo 9 weekly treatment sessions. The education group will receive learning materials about depression and will be monitored every month. All participants will have 4 study visits over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented as listed clinically in the participant's electronic medical record by any of the following tests: (1) any licensed rapid HIV test, (2) HIV enzyme test kit at any time prior to study entry, (3) at least one detectable HIV-1 antigen, or (4) at least one detectable plasma HIV-1 RNA viral load.
* Age ≥ 18 years.
* Ongoing receipt of stable antiretroviral therapy of any kind for at least 180 days prior to Screening
* Meets the depression definition for this trial:

  * (1) repeat PHQ-9 ≥10100 result at the Screening Visit (suggesting moderate to severe depressive symptoms), AND
  * (2) PHQ-9 depressive disorder diagnosis (2 or more of the 9 depressive symptoms, including depressed mood or anhedonia, present in the past 2 weeks), AND
  * (3) functional impairment (using the tenth PHQ-9 item assessing social/occupational impairment), AND
  * (4) no evidence that the direct physiological effects of a substance, medication, or medical condition clearly account for the depressive symptoms, AND
  * (5) no bipolar or psychotic disorders

NOTE: The use of antidepressant medications is not exclusionary.

* HbA1c < 6.5% at Screening
* HIV-1 RNA level < 75 copies/mL at Screening

NOTE: There are no CD4 cell count eligibility criteria for this trial.

Exclusion Criteria:

* Inability to complete written, informed consent
* Inability to read and understand English as seen on a computer screen
* Diagnosed diabetes mellitus or any previously recorded HbA1c ≥6.5%
* History of bipolar disorder or a psychotic disorder, including schizophrenia

NOTE: Depressive disorders are not exclusionary.

* Incarceration at the time of any study visit
* Active suicidality at Entry, as determined by the patient's HIV provider or social worker following a positive response (1, 2, or 3) to PHQ-9 Item #9 and a positive response (yes) to one or more of the three questions (for Question #3, the previous attempt must be within the past 10 years) on the Patient Suicidality Form (see Appendix).
* Diagnosed disease or process, besides HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosus, inflammatory bowel diseases, or other collagen vascular diseases).

NOTE: Hepatitis B or C co-infections are NOT exclusionary, but treatment for hepatitis C cannot be provided during study participation

* End stage renal disease requiring renal replacement therapy (dialysis, transplantation).
* Known or suspected malignancy requiring systemic treatment within 180 days of the Entry Visit.

NOTE: Localized treatment for skin cancers is not exclusionary.

• Therapy for serious medical illnesses within 14 days prior to the Entry Visit

NOTE: Therapy for serious medical illnesses that overlaps with a study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.

* Pregnancy or breastfeeding during the study.
* Receipt of investigational agents, cytotoxic chemotherapy, systemic immunosuppressive therapies, systemic glucocorticoids (of any dose), or anabolic steroids at the Entry Visit

NOTE: Physiologic testosterone replacement therapy or topical steroids is not exclusionary. Inhaled/nasal steroids are not exclusionary as long as the participant is not also receiving HIV protease inhibitors

NOTE: Use of NSAIDS and aspirin are allowed

• Active drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HOMA-IR at 24 weeks | 24 weeks
  Homeostasis Model Assessment-Insulin, where higher values indicate greater insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, Principal Investigator — Indiana University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Start date: January 1, 2031 End Date: Indefinite
Access Criteria: Data and sample requests will be honored after submission of a short proposal that outlines an important scientific question with an appropriate statistical analysis plan that justifies the use of these datasets. In addition, the requests must also verify that confidentiality of the datasets will be ensured. A formal data sharing agreement will be required prior to provision of any datasets.

REFERENCES:
- [Background] Bourgi K, Kundu S, Stewart JC, So-Armah K, Freiberg M, Gupta SK. Associations of HIV and Depression with Incident Diabetes Mellitus: Veterans Aging Cohort Study. Clin Infect Dis. 2022 Feb 3;78(2):378-85. doi: 10.1093/cid/ciac085. Online ahead of print. PMID 35134838
- [Background] Gupta SK, Slaven JE, Liu Z, Polanka BM, Freiberg MS, Stewart JC. Effects of Internet Cognitive-Behavioral Therapy on Depressive Symptoms and Surrogates of Cardiovascular Risk in Human Immunodeficiency Virus: A Pilot, Randomized, Controlled Trial. Open Forum Infect Dis. 2020 Jul 5;7(7):ofaa280. doi: 10.1093/ofid/ofaa280. eCollection 2020 Jul. PMID 32760749

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Version 1.0 updated Jan 27, 2026 (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT07226128/Prot_SAP_002.pdf
  • Informed Consent Form (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT07226128/ICF_003.pdf